CLINICAL TRIAL: NCT06865066
Title: Developing an Internet-Delivered Cognitive Behaviour Therapy Program for Women with Perimenopausal Anxiety: a Feasibility and Acceptability Study
Brief Title: Internet-Delivered Cognitive Behaviour Therapy for Women with Perimenopausal Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nazanin Alavi (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Principal Investigator, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6041810
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Menopause; Anxiety; Depressive/Anxiety Symptoms; Perimenopause
Keywords: Menopause; Anxiety; Online Psychotherapy; e-CBT; CBT; ACT; Menopause Transition; Digital Therapy; Perimenopause; Perimenopausal Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This one-arm trial will deliver e-CBT for perimenopausal anxiety using the Online Psychotherapy Tool (OPTT), a secure, cloud-based digital mental health platform. All participants will be enrolled in a 9-week e-CBT/e-ACT program specifically designed to address perimenopausal anxiety. Each week, they will complete structured e-modules and homework assignments while receiving personalized feedback and asynchronous support from a therapist through the platform. The program consists of 9 weekly sessions, each containing approximately 30 e-module slides with interactive content, all delivered through OPTT. This structured approach aims to help participants effectively manage their anxiety symptoms during perimenopause.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Online psychotherapy treatment arm (Experimental): All participants will receive access to e-CBT modules offered through the Online Psychotherapy Tool (OPTT) and will be paired with an online careprovider, who is trained to administer online CBT and ACT. Following the structure of previous e-CBT modules developed by the QUOPL team, the module for this study will be designed to mirror standard in-person CBT for Generalized Anxiety Disorder and will combine components of ACT. Weekly homework will be assigned and evaluated by the participant's designated care provider, who will provide personalized feedback on the online platform (OPTT), acknowledging their module completion and homework
  Interventions: Behavioral: e-CBT

INTERVENTIONS:
Behavioral: e-CBT — Electronically delivered cognitive behavioural therapy with acceptance commitment therapy components

SUMMARY:
The goal of this clinical trial is to design an online Cognitive Behavioural Therapy (CBT) and Acceptance Commitment Therapy (ACT) program and to learn if it can treat anxiety in women transitioning into menopause (perimenopause).

The main questions it aims to answer are:

* Is our online psychotherapy program a practical and acceptable means of managing anxiety during perimenopause?
* Does our online psychotherapy program work in improving anxiety levels during perimenopause?

Participants will participate in weekly e-CBT module sessions tailored to perimenopausal anxiety and will be given weekly feedback on assignments from trained care providers through a secure online platform. Participants will complete questionnaires at the beginning, middle, and at end of the study, as well as at the three and six-month follow-up.

DETAILED DESCRIPTION:
Participants (n=25) aged 40-60 years, experiencing perimenopause, as defined by the Stages of Reproductive Aging Workshop +10 (STRAW +10) criteria (a set of guidelines used to define the stages of early, late, and post-menopause, as indicated by hormone levels and change in menstrual activity) (Harlow et al., 2012), will be recruited from psychiatric and gynecology clinics at Kingston Health Sciences Centre (KHSC) and primary care providers in Kingston, ON. Study advertising will be conducted through social media advertisements, and flyers, which will be distributed to the email list of primary care providers in Kingston, ON and specialists (psychiatrists and gynecologists) at KHSC. This list has been compiled by QUOPL, which has developed it through research conducted in Kingston, ON over the past few years. Primary healthcare providers and specialists responsible for patient care in Kingston, ON and KHSC will assist in referring eligible patients to participate in the study. Referring healthcare providers will provide patients with flyers containing study information and clarify that, as their healthcare provider, they remain neutral regarding the patient's decision to participate.

If the patient wishes to proceed, they should contact the study coordinator whose contact information will be provided on the flyer. The coordinator will then arrange a virtual (Zoom) appointment with the patient to further discuss the study details and next steps. The letter of information will be emailed to the patient in advance and thoroughly reviewed during the Zoom meeting. Participants will be informed of their right to withdraw consent at any point, for any reason, without affecting their care or facing any consequences. If the patient still wishes to participate, they may provide verbal consent to proceed with the screening process. Upon receiving the patient's informed consent, the research coordinator will proceed with screening measures to confirm their eligibility. Subsequently, an appointment will be booked to confirm the diagnosis of Generalized Anxiety Disorder according to the Diagnostic And Statistical Manual Of Mental Disorders, Fifth Edition (DSM-5) criteria, utilizing the Mini International Psychiatric Assessment (MINI), English version 7.0.2 for DSM-5 by a trained research assistant.

During the meeting, the research coordinator will encourage participants to ask any questions they may have and will strive to provide thorough responses to the best of their ability. We will uphold strict confidentiality, refraining from disclosing any identifying information to anyone other than the study coordinator and the clinicians/physicians directly involved in the patient's care. All data collected from participants will be linked solely to their unique study ID. The study coordinator alone will possess the ability to connect the participant's ID with their name, which will be securely stored on a spreadsheet located on the QUOPL secure encrypted server. Other members of the study team will be granted access to de-identified participant data. All participants will receive a login to access their e-CBT modules offered through the Online Psychotherapy Tool (OPTT). OPTT is a secure, cloud-based digital mental health platform that complies with the Health Insurance Portability and Accountability Act, Personal Information Protection and Electronic Documents Act, and Service Organisation Control-2. In addition, all servers and databases are hosted in the Amazon Web Service Canada cloud infrastructure, which is managed by Medstack to ensure that all provincial and federal privacy and security regulations are met. OPTT does not collect any identifiable personal information or internet protocol addresses for privacy purposes. OPTT only collects anonymized metadata to improve its service quality and provide advanced analytics to the clinician team. OPTT encrypts all data, and no employees have direct access to participants' data. All encrypted backups are kept in the S3 storage that is dedicated to Queen's University, located in Kingston, Ontario, Canada.

Sessions will mirror the following weekly topics:

Session 1: What is Perimenopause and how can it Affect me?- Provides expectations for the course and introduces CBT and ACT in the context of perimenopause.

Session 2: Building a Foundation: Clarifying Values and Embracing Acceptance- Identifying symptoms of perimenopause and identifying risk factors (lifestyle, hormonal changes, changing work or familial roles) that may exacerbate symptoms. Upon onset, menopause carries on throughout a woman's life until post-menopausal staging. As such, some aspects of CBT (for example: experimentation) may not be well-suited or appropriate for menopause. In these instances, ACT will be introduced to teach situational acceptance and self-compassion. This session will explain how the first three strategies of ACT (Mindfulness, Values Clarification, and Cognitive Defusion) will be incorporated into CBT sessions throughout the course.

Session 3: Taking Action: Observing the Self and Committing to Change- This session teaches the last three ACT-based strategies for managing anxiety during perimenopause (Acceptance, Observing Self, Committed Action).

Session 4: The 5-part model for CBT (overview)- Introduces the concept of the 5-part Model and how situations, thoughts, feelings, physical reactions, and behaviours are connected and interact with each other.

Session 5: Situation, thoughts, feelings, physical reactions, and behaviours- Conceptualizes the 5 Part Model in detail, specifically how thoughts, feelings, behaviour, and physical reactions and one's environment interact and how changes in one area can affect the other 4 domains.

Session 6: The Thought Record- Highlights the first three columns of the Thought Record. The Thought record is a tool participants can use to dissect and understand the connection between feelings, behaviours, and thoughts. The first three columns include the situation, followed by the feelings and automatic thoughts associated with the situation. This session also discusses the role of automatic thoughts and how they influence feelings. The focus of this session is to understand how to identify automatic thoughts and specifically identify the most dominant idea, known as the "hot thought" when presented with a stressful situation. Common thinking distortions are also discussed in this session, as they apply to areas which may be relevant to perimenopause such as self-image, stigma, and managing symptoms in the workplace.

Session 7: Sleep Hygiene- Focuses on sleep habits with a particular focus on managing vasomotor symptoms at night. This session provides a variety of tips and strategies to use to increase sleep hygiene and get better quality rest.

Session 8: Evidence and Alternative & Balanced Thoughts- Focuses on the fourth and fifth columns of the Thought Record to help gather information that supports or does not support the identified hot thought. Also highlights the final sixth and seventh columns of the Thought Record which reflects on the evidence columns to help find an alternative or balanced view of the situation. The last column invites the participant to re-rate their feelings based on the completion of the Thought Record activity.

Session 9: Review & Maintenance- The final session is a review of the course and summarizes the main CBT and ACT concepts and tools that have been taught throughout the program and encourages users to continue using these skills beyond the transition to menopause.

Weekly homework will be assigned and evaluated by the participant's designated care provider, who will provide personalized feedback on OPTT, acknowledging their module completion and homework. Care providers will receive guidance in the form of sample feedback templates and scripts, serving as frameworks for optimizing interactions on the platform. These resources, drawn from previous research studies, will aid care providers in tailoring their services. To cater to individual participant needs, each session will feature a unique feedback template and script. These templates follow a standardized structure, commencing with recognition of the participant's progress. They also entail discussion of previously covered cognitive behavioural therapy (CBT) concepts, review of homework activities, validation of experiences, and encouragement to maintain attendance.

Participants will complete a series of validated questionnaires at five time points: at baseline (week 1), mid-point (week 4), post-treatment (week 9), and at the 3 and 6-month follow-up. These questionnaires are the Menopausal Rating Scale (MRS-II), Menopause-Specific Quality of Life Questionnaire (MENO-QOL), Perceived Stress Scale (PSS), Pittsburgh Sleep Quality Index (PSQI), General Anxiety-7 (GAD-7), Center for Epidemiologic Studies Depression Scale (CES-D), Depression Anxiety Stress Scale (DASS-21), and RAND 36-Item Short Form Health Survey (SF-36). At the beginning of the study, a demographic questionnaire will be administered. At the end of the study, a Qualtrics Survey will be administered to obtain general feedback on the program components.

Participants (n=8), including those who dropped out or were removed due to non-compliance at any stage of the study, will take part in a post-study interview led by a trained research assistant on the research study team. All interviews will be conducted in a semi-structured format following the study interview guide and will take place virtually via Zoom. The objective of the interview is to receive feedback regarding the relevance, effectiveness, and user-ease of this treatment program. In addition, the interview will provide insight into factors impacting their adherence and engagement throughout the study. An open-ended question guide will be used which focuses on patients' experiences. The interviewer may ask follow-up questions at their discretion to probe, obtain clarification, or expand on relevant topics that may not exactly follow the interview guide. The interviews will be approximately 40-60 minutes in length and will be recorded for transcription and coding purposes. A psychiatrist from the research team will be on-call during the virtual interview in case the patient needs extra support or is experiencing distress during the interviewing process. Should the patient be in crisis at any point during the interview, the interview will cease and the physician will be available to address the situation. In this context, crisis is defined as acute mental health symptoms that need attention. In cases of extreme crises where immediate care is needed, the research team will also call 9-1-1 (Emergency Telephone Number in Canada) or the crisis line on behalf of the patient.

ELIGIBILITY:
Inclusion Criteria:

* In perimenopausal staging (as defined by the STRAW +10 criteria)
* Assigned female at birth
* Diagnosis of GAD according to DSM-5 by attending psychiatrist on research team
* Competence to consent to participate
* Ability to speak and read English
* Consistent and reliable access to the internet

Exclusion Criteria:

* Undergone CBT or hormone therapy within the last 6 months will be excluded
* Active psychosis
* Acute mania
* Severe alcohol or substance use disorder
* Active suicidal or homicidal ideation

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms (Generalized Anxiety Disorder - 7 Item) | Week 0, week 4, week 9, 3 and 6-month follow-up
  Clinically validated symptom questionnaire. Scale of 0-3, 3 being the worst.

SECONDARY OUTCOMES:
Change in symptoms (Menopausal Rating Scale) | Week 0, week 4, week 9, 3 and 6-month follow-up
  Clinically validated symptom questionnaire. Scale of 0-4, 4 being the worst level of severity
Change in symptoms (Depression Anxiety Scale - 21 Item) | Week 0, week 4, week 9, 3 and 6-month follow-up
  Clinically validated symptom questionnaire. Scale of 0-3, 3 being the worst.
Change in symptoms (The Menopause-specific Quality of Life) | Week 0, week 4, week 9, 3 and 6-month follow-up
  Clinically validated symptom questionnaire. Scale of 0-6, 6 being the worst level of severity
Change in symptoms (Center for Epidemiologic Studies Depression Scale) | Week 0, week 4, week 9, 3 and 6-month follow-up
  Clinically validated symptom questionnaire. Scale of 0-3, 3 being the worst level of severity
Change in symptoms (Pittsburgh Sleep Quality Index) | Week 0, week 4, week 9, 3 and 6-month follow-up
  Clinically validated symptom questionnaire. Scale of 0-3, 3 being the worst.
Change in symptoms (Perceived Stress Scale) | Week 0, week 4, week 9, 3 and 6-month follow-up
  Clinically validated symptom questionnaire. Scale of 0-4, 4 being the worst level of severity.
Change in symptoms (RAND 36-Item Short Form Health Survey) | Week 0, week 4, week 9, 3 and 6-month follow-up
  Clinically validated symptom questionnaire assessing 8 domains with various scales.

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, MD, FRCPC, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - Nazanin Alavi, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No
Results will be shared through conference presentations, workshops, and journal publications.